CLINICAL TRIAL: NCT04452487
Title: Study of the Consequences of Infection on Compliance of Modalities of Decisions of Limitations and Stops of Treatments
Brief Title: Study of the Consequences of Infection on Compliance of Modalities of Decisions of Limitations and Stops of Treatments (COVID-19-LAT)
Acronym: COVID-19-LAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_GUASTELLA_COVID-19-LAT
Record Dates: First submitted 2020-06-23; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Patient Hospitalized in Disease Infectious Unit; Patient Hospitalized in Intensive Reanimation Unit; Patient Hopsitalized in Internal Medicine Unit
Keywords: COVID 19; Limitations and stops of processing Active Therapeutic; ethics; Sanitary Crisis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient 2019: Patients hospitalized in selected centers during march and june 2019
  Interventions: Behavioral: decisions of limitations and stop processing
- Patient 2020: Patients hospitalized in selected centers during march and june 2020 (during COVID-19 pandemia)
  Interventions: Behavioral: decisions of limitations and stop processing
- Patient 2021: Patients hospitalized in selected centers during march and june 2021
  Interventions: Behavioral: decisions of limitations and stop processing

INTERVENTIONS:
Behavioral: decisions of limitations and stop processing — Compliance of the modalities of decisions of limitations and stop processing

SUMMARY:
This survey is performed to examine if during the Covid's crisis, the practitionner's have respected the modalities of the law about the end of life, in particular concerning limitations and stop of therapeutics

DETAILED DESCRIPTION:
In the current legislativ context notably the Clayes Leonetti law, a very large majority of ICU (Intensive Care Unit) patients die with the establishement of a procedure for the limitation and cessation of therapeutics (LAT). During a viral pandemic, medical resources can be saturated, limiting reflexive abilities in favour of binary decisions. This sorting of patients leads to LAT that could be performed without the elementary modalities stated by the law. Thus, arbitrary medical decisions made alone could expose patients to unjustified " loss of luck ". Increasing the resources mobilized during a pandemic must not make us forget the quality of care provided for the benefit of quantity. In therefore seems legitimate to keep the LAT modalities to ensure our ethical principles. No work in the literature based on actual facts explores the impact of a pandemic on compliance with and maintenance of ethical principles and the legisltaive framework, in particular as regards the procedures of the application of LAT.

The purpose of this study is to assess whether the terms of the LAT are being complied during a pandemic for patients with or without Covid.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized major patient
* Infected or not with Covid-19
* having a management with a LAT defined by an anticipated or factual restriction of a therapeutic resource ( organ replacement, specific treatment) while his or her state of health requires or may require it, leading or not a death. The patient's death occurs either after a cariac massagewhich corresponds to a maximum management with therapeutic failure or within the framework or in the context of brain death, in these cases there is no LAT ; either without cardiac massage and in this case there is de facto a LAT wether or not it is performed according to legisltaive procedures. All patients who die will beclassified according to this diagram for the inclusion criterion. For surviving patients, an analysis of the record in search of LAT elments will be performed. In the absence of LAT elment in the record, i twill be considered that the patient did not have LAT and therfore will not be included.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in disease infectious Unit, or Patient hospitalized in intensive reanimation Unit, or Patient hopsitalized in Internal medicine Unit.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
decisions of limitations and therapeutic stops | at the end of patient's hospitalization, an average of one month
  The conformity of the modalities of the decisions of limitations and therapeutic stops will be evaluated by a composite criterion defined by the simultaneous presence of the 3 main modalities imposed by the Clayes-Leonetti law to achieve a limitation that are : An outside consultant's opinion ( required if no advance directives), the caregiver collegial discussion or adherence to patient advance directives, notification of decision in the medical record

SECONDARY OUTCOMES:
Characteristics of the notification of LAT procedure | at the end of patient's hospitalization, an average of one month
  notification of the decision, the conclusions of the discussions, the opinion of the consultant and the arguments given to justify the LAT
Characteristics of the LAT procedure (persons who participated to the collegial discussion) | at the end of patient's hospitalization, an average of one month
  number and status of caregivers who participated to the collegial discussion
Characteristics of consultant's reasoned opinion for the LAT procedure | at the end of patient's hospitalization, an average of one month
  formal elements of the consultant's reasoned opinion ( legal term) in the file
Characteristics of the LAT procedure | at the end of patient's hospitalization, an average of one month
  formal elements of advance directives
Characteristics of units | day 0
  number of beds, number of caregivers (medical, paramedical, internal external), number of admissions during periods of study
Age of physicians | Day 0
  measured in year
gendrer of physicians | Day 0
  male or female
Exparience of physicians | Day 0
  Measured in year of experience
Characteristics of physicians | Day 0
  professional status
Age of patients | day 0
  measured in year
patient's history | day 0
  comorbidities
COVID-19 patient's status | day 0
  COVID19 infection (yes or no)
Characteristics of hospitalization's patients | day 0
  hospitalization reason
Characteristics of affected organ | day 0
  organ failure
Characteristics of patients | day 0
  severity score
final patient status | day 0
  fate
patient's environnement | day 0
  family presence or relatives

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Guastella, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (3):
- France (3):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hospices Civiles de Lyon, Lyon
  - CH de Vichy, Vichy

REFERENCES:
- [Derived] Guastella V, Lambert C, Lafforgue A, Metretin P, Verstreate A, Watelet S, Perceau-Chambard E, Lautrette A. Withholding or withdrawing life-sustaining treatments in the COVID-19 pandemic: adherence to legal standards. BMJ Support Palliat Care. 2023 Aug 3:spcare-2023-004504. doi: 10.1136/spcare-2023-004504. Online ahead of print. PMID 37536752